CLINICAL TRIAL: NCT02499406
Title: Dialectical Behavior Therapy Skills Group Pilot Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Connecticut Healthcare System (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VACHS HSS 01883
Record Dates: First submitted 2015-06-01; First posted 2015-07-16 (Estimated); Results first posted 2020-01-02 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2020-01

CONDITIONS: Suicidal Ideation; Emotions
MeSH Terms: conditions — Suicidal Ideation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Skills group (Other): Dialectical behavior therapy skills group
  Interventions: Behavioral: Dialectical behavior therapy skills group

INTERVENTIONS:
Behavioral: Dialectical behavior therapy skills group — Skills training in emotion regulation, distress tolerance, interpersonal effectiveness, and mindfulness

SUMMARY:
Uncontrolled pilot study examines feasibility, acceptability, and preliminary efficacy of Dialectical Behavior Therapy skills group for Veterans with suicidal ideation and emotion dysregulation.

DETAILED DESCRIPTION:
Uncontrolled pilot study to examine feasibility, acceptability, and preliminary efficacy of Dialectical Behavior Therapy skills group for Veterans with suicidal ideation and emotion dysregulation. Outcome measures will occur at pre-treatment, mid, end, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Veterans at VACHS who are referred or self-referred to DBT Skills Group
2. Ages 18-65
3. Able to understand written and spoken English
4. DERS score 105 or greater
5. Suicidal ideation within past 3 months
6. Seeing an individual mental health provider at VACHS at least monthly
7. Willing to create or review a Mental Health Safety Plan, and stated willingness to use this plan to maintain safety
8. Consent to participate in study assessments
9. Consent to recording of group sessions

Exclusion Criteria:

1. Inability to understand written or spoken English
2. Diagnosis of schizophrenia, schizoaffective disorder, bipolar I, antisocial personality disorder, or thought disorder in CPRS problem list and confirmed by current mental health provider

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2014-12; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Decker, PhD, Principal Investigator — VA Connecticut Health Care System
Locations (1):
- VA Connecticut Health Care System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Skills Group
Started | 17
Completed | 13
Not Completed | 4
Not completed — missed 3 treatment sessions | 4

BASELINE CHARACTERISTICS:
Arm/Group | Skills Group
Number analyzed (Participants) | 17
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.7 (11.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 13
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 17

OUTCOME MEASURES:

1. Primary Outcome: Feasibility as Assessed by Attendance at Sessions for Duration of Intervention (Percent of Sessions Attended)
Description: Participation in skills group as assessed by attendance at sessions for duration of intervention (percent of sessions attended)
Time Frame: 6 months
Population: Percent of sessions attended
Measure: Mean (Full Range); unit: percentage of sessions attended
Arm/Group | Skills Group
Number analyzed (Participants) | 17
percentage of sessions attended | 66.4 [11.5 to 100.0]

2. Secondary Outcome: Acceptability as Assessed by Positive Feedback on Written Satisfaction Evaluations Completed by Participants at Mid-point of Intervention
Description: Acceptability to participants on the "Client Satisfaction Scale" created for this study. Participants rated group satisfaction on 11 items using 7point scale. Scale is scored by calculating mean of the 11 items. Scale range is 1-7. A higher score indicates greater satisfaction; a lower score indicates greater dissatisfaction, with 4 as the midpoint.
Time Frame: 3 months
Population: 17 participants started the study; 15 provided scores on this measure at 3-month assessment.
Measure: Mean (Standard Deviation); unit: score on a scale of satisfaction
Arm/Group | Skills Group
Number analyzed (Participants) | 15
score on a scale of satisfaction | 5.44 (0.50)

3. Secondary Outcome: Acceptability as Assessed by Positive Feedback on Written Satisfaction Evaluations Completed by Participants at Post-intervention
Description: as for outcome 2
Time Frame: 6 months
Population: 17 participants started the study; 12 provided scores on this measure at 6-month assessment.
Measure: Mean (Standard Deviation); unit: score on a scale of satisfaction
Arm/Group | Skills Group
Number analyzed (Participants) | 12
score on a scale of satisfaction | 6.17 (0.50)

4. Secondary Outcome: Acceptability as Assessed by Positive Feedback on Written Satisfaction Evaluations Completed by Participants at Follow-up
Description: as for outcome 2
Time Frame: 9 months
Population: 17 participants started the study; 12 provided scores on this measure at 9-month assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills Group
Number analyzed (Participants) | 12
score on a scale | 5.97 (0.39)

5. Secondary Outcome: Suicidal Ideation on Suicidal Behavior Questionnaire at 3months
Description: Scale title: Suicidal Behavior Questionnaire. Minimum value = 0, maximum value = 92. Higher score indicates greater suicidal ideation; lower score indicates lower suicidal ideation.
Time Frame: 3 months
Population: 17 participants started the study; 15 provided scores on this measure at 3month assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills Group
Number analyzed (Participants) | 15
score on a scale | 38.47 (15.43)
Statistical Analysis 1: Comparison: Skills Group; Null hypothesis is that there is no difference between baseline assessment and this 3-month assessment; Test type: Superiority; p > 0.016, paired sample t-test — a priori threshold for significance adjusted to p = .016 for multiple comparisons; df=14

6. Secondary Outcome: Suicidal Ideation on Suicidal Behavior Questionnaire at 6months
Description: as for outcome 5
Time Frame: 6 months
Population: 17 participants started the study. 12 contributed data on this measure at 6month assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills Group
Number analyzed (Participants) | 12
score on a scale | 29.00 (22.19)
Statistical Analysis 1: Comparison: Skills Group; Null hypothesis is that there is no difference between baseline assessment and this 6-month assessment; Test type: Superiority; p < 0.016, paired sample t-test — p value was calculated and found to be below the a priori threshold for significance, which was adjusted to p = .016 for multiple comparisons; df=11

7. Secondary Outcome: Suicidal Ideation on Suicidal Behavior Questionnaire at 9months
Description: as for outcome 5
Time Frame: 9 months
Population: 17 participants started the study. 12 contributed data on SBQ at 9month assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills Group
Number analyzed (Participants) | 12
score on a scale | 28.25 (19.81)
Statistical Analysis 1: Comparison: Skills Group; Null hypothesis is that there is no difference between baseline assessment and this 9-month assessment; Test type: Superiority; p < 0.016, paired sample t-test — a priori threshold for significance adjusted to p = .016 for multiple comparisons; df=11

8. Secondary Outcome: Emotion Dysregulation as Assessed Using Difficulties in Emotion Regulation Scale at 3months
Description: Scale title: Difficulties in Emotion Regulation Scale (DERS). Scale range: 36-180. Higher score indicates greater difficulties regulating emotions. Lower score indicates fewer difficulties regulating emotions.
Time Frame: 3 months
Population: 17 participants started the study; 15 provided data on this measure at 3months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills Group
Number analyzed (Participants) | 15
score on a scale | 107.27 (15.20)
Statistical Analysis 1: Comparison: Skills Group; Null hypothesis is that there is no difference in paired samples between baseline and 3-month assessment; Test type: Superiority; p < 0.016, paired samples t test — a priori threshold for significance adjusted to p = .016 for multiple comparisons; df=14

9. Secondary Outcome: Emotion Dysregulation as Assessed Using Difficulties in Emotion Regulation Scale at 6months (End of Intervention)
Description: as for outcome 8
Time Frame: 6 months
Population: 17 participants started the study. 11 contributed data on DERS at 6months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills Group
Number analyzed (Participants) | 11
score on a scale | 86.27 (12.81)
Statistical Analysis 1: Comparison: Skills Group; Null hypothesis is no difference between baseline and this 6-month assessment; Test type: Superiority; p < 0.016, paired samples t test — a priori threshold for significance adjusted to p = .016 for multiple comparisons; df=10

10. Secondary Outcome: Emotion Dysregulation as Assessed Using Difficulties in Emotion Regulation Scale at 9months
Description: as for outcome 8
Time Frame: 9 months
Population: 17 participants started the study. 12 contributed data on DERS at 9months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills Group
Number analyzed (Participants) | 12
score on a scale | 84.92 (15.31)
Statistical Analysis 1: Comparison: Skills Group; Null hypothesis is no difference between baseline and this 9-month assessment; Test type: Superiority; p < 0.016, paired samples t test — a priori threshold for significance adjusted to p = .016 for multiple comparisons; df=11

11. Secondary Outcome: Coping as Assessed With the DBT (Dialectical Behavior Therapy) Ways of Coping Checklist at 3months
Description: Scale title: Dialectical Behavior Therapy Ways of Coping Checklist (DBT-WCCL) effective coping subscale. Minimum score: 0. Maximum score: 3. Higher score indicates more frequent use of adaptive coping strategies. Lower score indicates less frequent use of adaptive coping strategies.
Time Frame: 3 months
Population: 17 participants started the study. 15 contributed data on this measure at 3 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills Group
Number analyzed (Participants) | 15
score on a scale | 1.51 (0.40)
Statistical Analysis 1: Comparison: Skills Group; Null hypothesis is that there is no difference between baseline assessment and this 3-month assessment; Test type: Superiority; p > 0.016, paired sample t test — a priori threshold for significance adjusted to p = .016 for multiple comparisons; df=14

12. Secondary Outcome: Coping as Assessed With the DBT Ways of Coping Checklist at 6 Months
Description: as for outcome 11
Time Frame: 6 months
Population: 17 participants started the study. 11 participants contributed data on this measure at 6month assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills Group
Number analyzed (Participants) | 11
score on a scale | 1.80 (0.41)
Statistical Analysis 1: Comparison: Skills Group; Null hypothesis is that there is no difference between baseline assessment and this 6-month assessment; Test type: Superiority; p = .016, paired sample t-test — a priori threshold for significance adjusted to p = .016 for multiple comparisons; df=10

13. Secondary Outcome: Coping as Assessed With the DBT Ways of Coping Checklist at 9months
Description: as for outcome 11
Time Frame: 9 months
Population: 17 participants started the study; 12 contributed data on this measure at 9months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Skills Group
Number analyzed (Participants) | 12
score on a scale | 1.83 (0.50)
Statistical Analysis 1: Comparison: Skills Group; Null hypothesis is that there is no difference between baseline assessment and this 9-month assessment; Test type: Superiority; p < 0.016, paired sample t-test — a priori threshold for significance adjusted to p = .016 for multiple comparisons; df=11

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Skills Group
All-Cause Mortality (participants affected / at risk) | 0/17
Serious Adverse Events (participants affected / at risk) | 1/17
Other Adverse Events (participants affected / at risk) | 0/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Skills Group (N=17)
inpatient hospitalization (Psychiatric disorders) | 1 (1) — psychiatric hospitalization in a participant who had previously dropped out of study

LIMITATIONS AND CAVEATS:
Some missing data in assessments due to attrition; planned absence of control arm for this small open feasibility pilot trial; absence of adherence coding due to logistical constraints

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT02499406/Prot_SAP_000.pdf